CLINICAL TRIAL: NCT00602225
Title: Dose Escalation Study of Clofarabine in Combination With Cytarabine (Ara-C) and G-CSF Priming for Relapsed or Refractory Acute Myeloid Leukemia (AML) Patients
Brief Title: Clofarabine, Cytarabine, and G-CSF in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela S Becker, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6562; NCI-2009-01464 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Acute Myeloid Leukemia; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Promyelocytic Leukemia (M3); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Promyelocytic, Acute | interventions — Clofarabine; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Drug: clofarabine; Drug: cytarabine; Biological: filgrastim

INTERVENTIONS:
Drug: clofarabine — Given IV
  Other Names: CAFdA; Clofarex; Clolar
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Biological: filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or stopping them from dividing. Colony stimulating factors, such as G-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy.

PURPOSE: This phase I trial is studying the side effects and best dose of clofarabine to see how well it works when given together with cytarabine and G-CSF in treating patients with relapsed or refractory acute myeloid leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of clofarabine, and the dose-limiting toxicities of the combination of clofarabine and cytarabine with G-CSF priming, in the treatment of patients with relapsed or refractory AML.

SECONDARY OBJECTIVES:

I. To determine the hematological and non-hematological side effect profile of the combination of clofarabine, cytarabine, and G-CSF.

II. To determine the efficacy of clofarabine in combination with cytarabine and G-CSF priming in the treatment of patients with relapsed or refractory AML.

III. To determine the disease-free and overall survival after therapy with clofarabine, cytarabine, and G-CSF for relapsed or refractory AML.

OUTLINE: This is a dose escalation study of clofarabine.

PART I:

INDUCTION THERAPY: Patients receive clofarabine IV over 1 hour and cytarabine IV over 2 hours on days 1-5, and filgrastim (G-CSF) subcutaneously once daily beginning 24 hours prior to chemotherapy and continuing until blood count recover. Patients with residual leukemia (>= 5% blasts by morphology) at day 14 and if blast remain > 5% by day 21 receive a second course of induction therapy.

CONSOLIDATION THERAPY: Patients receive clofarabine, cytarabine, and G-CSF as in induction therapy. Patients may receive a second course of consolidation therapy depending on response and whether additional therapy (e.g., stem cell transplant or donor lymphocyte infusion) is planned.

PARTS II and III:

Patients receive induction therapy and consolidation therapy as in part 1.

After completion of study treatment, patients are followed every 3 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female patients must be willing to use an effective contraceptive method during the study and for a minimum of 6 months after study treatment
* Serum Total or Direct bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2.5 times ULN
* Diagnosis of acute myeloid leukemia by WHO criteria, either relapsed or refractory; acute promyelocytic leukemia [acute promyelocytic leukemia with t(15;17)(q22;q12) and variants] would be eligible only after failure of a regimen containing arsenic trioxide
* Serum creatinine =< 1.0 mg/dL; if serum creatinine > 1.0 mg/dl, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m^2
* Alkaline phosphatase =< 2.5 times ULN

Exclusion Criteria:

* Use of investigational agents within 30 days or initiation of any other anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea, and intrathecal therapy for leukemic meningitis
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Have any other severe concurrent disease, history of serious organ dysfunction, or disease involving the heart, kidney, liver (including symptomatic hepatitis, veno-occlusive disease, or hepatic graft-versus-host disease [for acute >= grade 2]), or other organ system dysfunction
* No concomitant cytotoxic therapy or investigational therapy is allowed during the study with the exception of intrathecal therapy for leukemic meningitis; intrathecal therapy must not be given during or within 24 hours of any 5 day Clofarabine/Cytarabine treatment period
* To the extent possible, use of nephrotoxic (e.g., vancomycin, amphotericin B, etc) and hepatotoxic (e.g., voriconazole, cyclosporine, etc) agents is to be avoided during clofarabine; use of alternative medications (e.g., herbal or botanical for anticancer purposes) is not permitted during the entire study period
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* More than two failed induction attempts for initial diagnosis or current relapse; for patients enrolled under part III of the protocol, patients must be at first salvage after relapse less than one year from complete remission, or salvage after initial induction chemotherapy
* Allogeneic transplant recipients on immunosuppression or on treatment for GVHD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Becker, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Becker PS, Kantarjian HM, Appelbaum FR, Storer B, Pierce S, Shan J, Faderl S, Estey EH. Retrospective comparison of clofarabine versus fludarabine in combination with high-dose cytarabine with or without granulocyte colony-stimulating factor as salvage therapies for acute myeloid leukemia. Haematologica. 2013 Jan;98(1):114-8. doi: 10.3324/haematol.2012.063438. Epub 2012 Jul 16. PMID 22801963

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Filgrastim + Clofarabine + Cytarabine (GCLAC): See Detailed Description
  clofarabine: Given IV
  cytarabine: Given IV
  filgrastim: Given subcutaneously
Period: Overall Study
Arm/Group | Arm I: Filgrastim + Clofarabine + Cytarabine (GCLAC)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 53 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 36
AML Onset: de novo [Count of Participants; unit: Participants] — Number of participants whose diagnosis of Acute Myeloid Leukemia was not preceded by an Antecedent Hematological Disorder or treatment with chemotherapy/radiation.
  Participants | 32
AML Onset: secondary [Count of Participants; unit: Participants] — Number of participants whose diagnosis of Acute Myeloid Leukemia was preceded by an Antecedent Hematological Disorder or treatment with chemotherapy/radiation.
  Participants | 18
Relapsed [Count of Participants; unit: Participants] — Number of patients with relapsed Acute Myeloid Leukemia
  Participants | 32
First salvage [Count of Participants; unit: Participants] — Number of participants for whom treatment on this protocol was considered first salvage therapy.
  Participants | 32
Second or greater salvage [Count of Participants; unit: Participants] — Number of participants for whom treatment on this protocol was considered second or greater salvage therapy.
  Participants | 18
Refractory [Count of Participants; unit: Participants] — Number of participants whose disease was considered refractory at the time of enrollment.
  Participants | 18
Favorable cytogenetics (at initial diagnosis) [Count of Participants; unit: Participants] — Number of participants who had favorable risk cytogenetics at initial diagnosis.
  Participants | 3
Intermediate cytogenetics (at initial diagnosis) [Count of Participants; unit: Participants] — Number of participants who had intermediate risk cytogenetics at initial diagnosis.
  Participants | 27
Unfavorable cytogenetics (at initial diagnosis) [Count of Participants; unit: Participants] — Number of participants who had unfavorable risk cytogenetics at initial diagnosis.
  Participants | 20
Median first CR duration [Median (Full Range); unit: weeks] — Population: This baseline measure only applies to those participants whose disease was in relapse at the time of enrollment.
  weeks
    number analyzed (Participants) | 32
    (all) | 26 [0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Clofarabine
Time Frame: 45 days after the last dose of clofarabine
Measure: Number; unit: mg/m^2 of clofarabine
Arm/Group | Arm I: Filgrastim + Clofarabine + Cytarabine (GCLAC)
Number analyzed (Participants) | 50
mg/m^2 of clofarabine | 25

2. Primary Outcome: Dose-limiting Toxicity as Assessed by NCI CTCAE v3.0
Time Frame: 45 days after the last dose of clofarabine
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Filgrastim + Clofarabine + Cytarabine (GCLAC)
Number analyzed (Participants) | 50
Participants | 2

3. Primary Outcome: Response Rates by Cytogenetic Risk Category
Description: Number of participants who achieved Complete Remission (less than 5% blasts in the marrow and count recovery of Absolute Neutrophil Count to 1,000/microL and Platelet Count to 100,000/microL) under each cytogenetic risk category.
Time Frame: 45 days after the last dose of clofarabine
Population: Of the 50 patients, 4 were excluded from analysis of response: 2 patients with GVHD, 1 patient who received only 1 g/m2 ara-C, and 1 patient who did not have a marrow confirming remission status prior to beginning a preparative regimen for allogeneic HCT.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 46
Participants
  Favorable risk Complete Remission: number analyzed (Participants) | 3
  Favorable risk Complete Remission | 3
  Intermediate risk Complete remission: number analyzed (Participants) | 25
  Intermediate risk Complete remission | 10
  Unfavorable risk Complete remission: number analyzed (Participants) | 18
  Unfavorable risk Complete remission | 9

4. Primary Outcome: Response Rates by Cytogenetic Risk Category and Clofarabine Dose
Description: Number of participants under each Cytogenetic Risk Category and Clofarabine dose who achieve CR (Complete Remission = less than 5% blasts in the marrow and count recovery of Absolute Neutrophil Count to 1,000/microL and Platelet Count to 100,000/microL) or CRp (Complete Remission, but with a platelet count of less than 100,000/microL).
Time Frame: 45 days after the last dose of clofarabine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 46
Participants
  Favorable Risk + 25 mg/m^2 achieve CR: number analyzed (Participants) | 3
  Favorable Risk + 25 mg/m^2 achieve CR | 2
  Intermediate Risk + 15 mg/m^2 achieve CR: number analyzed (Participants) | 4
  Intermediate Risk + 15 mg/m^2 achieve CR | 2
  Intermediate Risk + 20 mg/m^2 achieve CR: number analyzed (Participants) | 4
  Intermediate Risk + 20 mg/m^2 achieve CR | 3
  Intermediate Risk + 25 mg/m^2 achieve CR: number analyzed (Participants) | 17
  Intermediate Risk + 25 mg/m^2 achieve CR | 5
  Intermediate Risk + 25 mg/m^2 achieve CRp: number analyzed (Participants) | 17
  Intermediate Risk + 25 mg/m^2 achieve CRp | 4
  Unfavorable Risk + 15 mg/m^2 achieve CR: number analyzed (Participants) | 4
  Unfavorable Risk + 15 mg/m^2 achieve CR | 2
  Unfavorable Risk + 20 mg/m^2 achieve CR: number analyzed (Participants) | 2
  Unfavorable Risk + 20 mg/m^2 achieve CR | 1
  Unfavorable Risk + 25 mg/m^2 achieve CR: number analyzed (Participants) | 12
  Unfavorable Risk + 25 mg/m^2 achieve CR | 6
  Unfavorable Risk + 25 mg/mg^2 achieve CRp: number analyzed (Participants) | 12
  Unfavorable Risk + 25 mg/mg^2 achieve CRp | 3

5. Primary Outcome: Response Rates by Duration First Complete Remission (CR1)
Description: Number of participants whose first Complete Remission lasted 0, 1-6, 6-12, or greater than 12 months. Only those participant who had a first CR are included in this data.
Time Frame: 45 days after the last dose of clofarabine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 21
Participants
  Duration CR1 (months): 0 | 12
  Duration CR1 (months): 1-6 | 4
  Duration CR1 (months): 6-12 | 2
  Duration CR1 (months): greater than 12 | 3

6. Primary Outcome: Response Rates by Salvage Number
Description: Number of participants in each Salvage number category who achieved a Complete Remission. Salvage number refers to whether treatment with GCLAC on this study was the pariticipant's first salvage regimen (1), second salvage regimen (2), or third or greater salvage regimen (3 or greater).
Time Frame: 45 days after the last dose of clofarabine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 46
Participants
  Salvage number 1: number analyzed (Participants) | 33
  Salvage number 1 | 16
  Salvage number 2: number analyzed (Participants) | 8
  Salvage number 2 | 5
  Salvage number 3 or greater: number analyzed (Participants) | 5
  Salvage number 3 or greater | 0

7. Secondary Outcome: Hematologic and Non-hematologic Side Effect Profile
Time Frame: 45 days after the last dose of clofarabine
Population: Data not collected
Arm/Group | Arm I: Filgrastim + Clofarabine + Cytarabine (GCLAC)
Number analyzed (Participants) | 0

8. Secondary Outcome: Efficacy
Description: Number of Patients Surviving at Five Years
Time Frame: At five years after the last dose of clofarabine
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Filgrastim + Clofarabine + Cytarabine (GCLAC)
Number analyzed (Participants) | 50
Participants | 12

9. Secondary Outcome: Disease-free Survival
Description: Number of participants who survived and were disease-free at 5 years
Time Frame: At five years after the last dose of clofarabine
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Filgrastim + Clofarabine + Cytarabine (GCLAC)
Number analyzed (Participants) | 50
Participants | 11

10. Secondary Outcome: Overall Survival
Time Frame: At five years after the last dose of clofarabine
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 50
months | 9 [5.2 to 13]

ADVERSE EVENTS:
Description: Other [Non-serious] adverse events were not collected/assessed.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 23/50
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=50)
Skin (Skin and subcutaneous tissue disorders) | 5 (5)
Hepatic transaminases (Hepatobiliary disorders) | 8 (8)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 23 (23)
infection (Infections and infestations) | 20 (20)
Gastrointestinal (Gastrointestinal disorders) | 6 (6)
Hyperbilirubinaemia (Investigations) | 4 (4)
Renal (Renal and urinary disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Tumor Lysis (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No